CLINICAL TRIAL: NCT01788046
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Assess the Efficacy and Safety of AMG 416 in the Treatment of Secondary Hyperparathyroidism in Subjects With Chronic Kidney Disease on Hemodialysis
Brief Title: Efficacy and Safety of Etelcalcetide (AMG 416) in the Treatment of Secondary Hyperparathyroidism (SHPT) in Patients With Chronic Kidney Disease (CKD) on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120230; KAI-4169-007 (Other: KAI Pharmaceuticals, Inc (wholly owned subsidiary of Amgen Inc.)); 2012-002806-31 (EudraCT Number)
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: Secondary Hyperparathyroidism (SHPT), chronic kidney disease (CKD), hemodialysis, parathyroid hormone (PTH), hypocalcemia, bone and mineral metabolism
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Hypocalcemia | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo administered by intravenous bolus injection at the end of each hemodialysis session, three times per week (TIW) for 26 weeks.
  Interventions: Drug: Placebo
- Etelcalcetide (Experimental): Participants received etelcalcetide administered by intravenous bolus injection at the end of each hemodialysis session TIW for 26 weeks.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Administered intravenously three times per week. The starting dose was 5 mg. The dose may have been increased at weeks 5, 9, 13, and 17 (4-week intervals) by 2.5 mg or 5 mg on the basis of the predialysis parathyroid hormone and corrected calcium concentrations obtained in the prior week. The minimum dose was 2.5 mg and the maximum dose was 15 mg.
  Other Names: AMG 416
  Arms: Etelcalcetide
Drug: Placebo — Administered intravenously (IV) three times per week.
  Arms: Placebo

SUMMARY:
This study is designed to assess the efficacy and safety of etelcalcetide (AMG 416) compared with placebo in the treatment of SHPT in CKD patients receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
* Subject is 18 years of age or older.
* Subject agrees to not participate in another study of an investigational agent during the study.
* Subject must be receiving hemodialysis 3 times weekly for at least 3 months
* Other Inclusion Criteria may apply

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study, or ended treatment on another investigational device or drug study(s) within 8 weeks prior to screening.
* Other investigational procedures while participating in this study are excluded.
* Anticipated or scheduled parathyroidectomy during the study period.
* Subject has received a parathyroidectomy within 3 months prior to dosing.
* Anticipated or scheduled kidney transplant during the study period.
* Subject has known sensitivity to any of the products or components to be administered during dosing.
* Subject has participated in a prior clinical trial of AMG 416
* Subject has an unstable medical condition based on medical history, physical examination, and routine laboratory tests, or is otherwise unstable in the judgment of the Investigator.
* Subject has a history of any illness that, in the opinion of the Investigator, might confound the results of the study or pose additional risk to the subject.
* Other Exclusion Criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2014-04-14 (Actual); Study Completion 2014-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (102):
- United States (45):
  - Research Site, Mobile, Alabama
  - Research Site, Azusa, California
  - Research Site, Beverly Hills, California
  - Research Site, Chula Vista, California
  - Research Site, Fairfield, California
  - Research Site, Glendale, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Norwalk, California
  - Research Site, Riverside, California
  - Research Site, Simi Valley, California
  - Research Site, Denver, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Merrillville, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Ft. Washington, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Brookhaven, Mississippi
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Eatontown, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Fresh Meadows, New York
  - Research Site, Great Neck, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbia, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Rutland, Vermont
  - Research Site, Alexandria, Virginia
  - Research Site, Morgantown, West Virginia
- Australia (4):
  - Research Site, Westmead, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Clayton, Victoria
- Belgium (5):
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Liège
  - Research Site, Roeselare
  - Research Site, Tournai
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, New Westminster, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (4):
  - Research Site, Nový Jičín
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Ústí nad Orlicí
- France (5):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Grenoble
  - Research Site, Marseille
  - Research Site, Perpignan
- Research Site, Erfurt, Germany
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Esztergom
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Zalaegerszeg
- Israel (4):
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Tel Litwinsky
  - Research Site, Ẕerifin
- Italy (4):
  - Research Site, Ancona
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Quartu Sant'Elena CA
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Enschede
  - Research Site, Rotterdam
  - Research Site, Venlo
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Golub-Dobrzyń
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Rybnik
  - Research Site, Warsaw
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Spain (4):
  - Research Site, Córdoba, Andalusia
  - Research Site, Granada, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, Majadahonda, Madrid
- Sweden (3):
  - Research Site, Karlstad
  - Research Site, Stockholm
  - Research Site, Uppsala

REFERENCES:
- [Background] Block GA, Bushinsky DA, Cunningham J, Drueke TB, Ketteler M, Kewalramani R, Martin KJ, Mix TC, Moe SM, Patel UD, Silver J, Spiegel DM, Sterling L, Walsh L, Chertow GM. Effect of Etelcalcetide vs Placebo on Serum Parathyroid Hormone in Patients Receiving Hemodialysis With Secondary Hyperparathyroidism: Two Randomized Clinical Trials. JAMA. 2017 Jan 10;317(2):146-155. doi: 10.1001/jama.2016.19456. PMID 28097355
- [Background] Kroenke MA, Weeraratne DK, Deng H, Sloey B, Subramanian R, Wu B, Serenko M, Hock MB. Clinical immunogenicity of the d-amino acid peptide therapeutic etelcalcetide: Method development challenges and anti-drug antibody clinical impact assessments. J Immunol Methods. 2017 Jun;445:37-44. doi: 10.1016/j.jim.2017.03.005. Epub 2017 Mar 6. PMID 28274835
- [Background] Stollenwerk B, Iannazzo S, Akehurst R, Adena M, Briggs A, Dehmel B, Parfrey P, Belozeroff V. A Decision-Analytic Model to Assess the Cost-Effectiveness of Etelcalcetide vs. Cinacalcet. Pharmacoeconomics. 2018 May;36(5):603-612. doi: 10.1007/s40273-017-0605-2. PMID 29392552
- [Background] Stollenwerk B, Iannazzo S, Cooper K, Belozeroff V. Exploring the potential value of improved care for secondary hyperparathyroidism with a novel calcimimetic therapy. J Med Econ. 2017 Oct;20(10):1110-1115. doi: 10.1080/13696998.2017.1360309. Epub 2017 Aug 14. PMID 28803497
- [Background] Chen P, Narayanan A, Wu B, Gisleskog PO, Gibbs JP, Chow AT, Melhem M. Population Pharmacokinetic and Pharmacodynamic Modeling of Etelcalcetide in Patients with Chronic Kidney Disease and Secondary Hyperparathyroidism Receiving Hemodialysis. Clin Pharmacokinet. 2018 Jan;57(1):71-85. doi: 10.1007/s40262-017-0550-4. PMID 28508378
- [Background] Block GA, Chertow GM, Sullivan JT, Deng H, Mather O, Tomlin H, Serenko M. An integrated analysis of safety and tolerability of etelcalcetide in patients receiving hemodialysis with secondary hyperparathyroidism. PLoS One. 2019 Mar 15;14(3):e0213774. doi: 10.1371/journal.pone.0213774. eCollection 2019. PMID 30875390
- [Background] Cunningham J, Block GA, Chertow GM, Cooper K, Evenepoel P, Iles J, Sun Y, Urena-Torres P, Bushinsky DA. Etelcalcetide Is Effective at All Levels of Severity of Secondary Hyperparathyroidism in Hemodialysis Patients. Kidney Int Rep. 2019 Apr 16;4(7):987-994. doi: 10.1016/j.ekir.2019.04.010. eCollection 2019 Jul. PMID 31317120
- [Background] Wolf M, Block GA, Chertow GM, Cooper K, Fouqueray B, Moe SM, Sun Y, Tomlin H, Vervloet M, Oberbauer R. Effects of etelcalcetide on fibroblast growth factor 23 in patients with secondary hyperparathyroidism receiving hemodialysis. Clin Kidney J. 2019 Apr 26;13(1):75-84. doi: 10.1093/ckj/sfz034. eCollection 2020 Feb. PMID 32082556
- [Background] Hain D, Tomlin H, Gibson C. Administration of Etelcalcetide for the Treatment of Secondary Hyperparathyroidism in Patients with CKD-MBD on Hemodialysis: A Nephrology Nursing Perspective. Nephrol Nurs J. 2019 May-Jun;46(3):315-290. PMID 31199098
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 97 centers in the US, Canada, Europe, Israel, the Russian Federation, and Australia. The first participant was enrolled on 12 March 2013, and the last participant 07 October 2013.
Pre-assignment Details: Eligible participants were randomized 1:1 to etelcalcetide or placebo. Randomization was stratified by screening parathyroid hormone (PTH) (< 600 pg/mL, 600 to ≤ 1000 pg/mL, and > 1000 pg/mL), prior cinacalcet use and region (North America or non-North America).
Period: Overall Study
Arm/Group | Placebo | Etelcalcetide
Started | 260 | 255
Received Treatment | 259 | 252
Completed | 204 | 218
Not Completed | 56 | 37
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Lost to Follow-up | 12 | 19
Not completed — Death | 7 | 5
Not completed — Protocol Specified Criteria | 25 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Etelcalcetide | Total
Number analyzed (Participants) | 260 | 255 | 515
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (13.9) | 58.4 (14.6) | 58.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 93 | 188
  Male | 165 | 162 | 327
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 13 | 19
  Black (or African American) | 80 | 64 | 144
  Native Hawaiian or Other Pacific Islander | 3 | 7 | 10
  White | 169 | 163 | 332
  Other | 2 | 6 | 8
  Missing | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 33 | 32 | 65
  Not Hispanic/Latino | 227 | 221 | 448
  Missing | 0 | 2 | 2
Stratification Factor: Screening Serum Parathroid Hormone [Number; unit: participants]
  < 600 pg/mL | 84 | 84 | 168
  ≥ 600 to ≤ 1000 pg/mL | 121 | 118 | 239
  > 1000 pg/mL | 55 | 53 | 108
Stratification Factor: Cinacalcet Use Within 8 Weeks of Randomization [Number; unit: participants]
  Yes | 33 | 29 | 62
  No | 227 | 226 | 453
Stratification Factor: Region [Number; unit: participants]
  North America | 150 | 146 | 296
  Non-North America | 110 | 109 | 219
Parathyroid Hormone [Mean (Standard Deviation); unit: pg/mL] | 851.7 (552.0) | 845.0 (464.3) | 848.4 (510.0)
Phosphorus [Mean (Standard Deviation); unit: mg/dL] — Data available for 257 and 251 participants in each treatment group respectively
  mg/dL | 5.83 (1.45) | 5.76 (1.60) | 5.79 (1.53)
Corrected Calcium (cCa) [Mean (Standard Deviation); unit: mg/dL] | 9.70 (0.69) | 9.63 (0.65) | 9.66 (0.67)
Corrected Calcium Phosphorus Product (cCa x P) [Mean (Standard Deviation); unit: mg²/dL²] — Data available for 257 and 251 participants in each treatment group respectively
  mg²/dL² | 56.37 (14.50) | 55.30 (15.27) | 55.84 (14.88)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With > 30% Decrease From Baseline in Mean PTH During the Efficacy Assessment Phase
Description: Participants who did not have any scheduled assessments during the EAP were considered non-responders.
Time Frame: Baseline and the efficacy assessment phase (EAP; defined as Weeks 20 to 27, inclusive).
Population: The full analysis set, consisting of all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 260 | 255
percentage of participants | 9.6 | 75.3
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; A Cochran-Mantel-Haenszel test stratified by screening PTH category (< 600, ≥ 600 to ≤ 1000, and > 1000 pg/mL), recent cinacalcet use within 8 weeks before randomization (yes and no), and region (North America and non-North America) was used to compare the primary endpoint of percentage of participants with > 30% reduction from baseline in PTH during the EAP between etelcalcetide and placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 30.80, 95% CI 2-sided [18.18 to 52.17]

2. Secondary Outcome: Percentage of Participants With Mean Predialysis Parathyroid Hormone ≤ 300 pg/mL During the Efficacy Assessment Phase
Description: Participants who had no scheduled assessments during the EAP were considered non-responders.
Time Frame: Baseline and the efficacy assessment phase (Week 20 to Week 27)
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 260 | 255
percentage of participants | 4.6 | 53.3
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by screening PTH category, prior cinacalcet use within 8 weeks prior to randomization, and region; Odds Ratio (OR) = 33.92, 95% CI 2-sided [16.35 to 70.37]

3. Secondary Outcome: Percent Change From Baseline in Predialysis PTH During the Efficacy Assessment Phase
Time Frame: Baseline and the Efficacy Assessment Phase (Week 20 to Week 27)
Population: Full analysis set participants with observed data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 237 | 227
percent change | 13.72 (2.50) | -57.39 (1.91)
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p < 0.001, Repeated Measures Mixed Effects Model; Repeated measures mixed-effects model included treatment, stratification factors, visit, and treatment by visit interaction as covariates; Mean Difference = -71.34, 95% CI 2-sided [-77.53 to -65.14], Standard Error of Mean 3.15 — Etelcalcetide - Placebo

4. Secondary Outcome: Percent Change From Baseline in Predialysis Corrected Calcium During the Efficacy Assessment Phase
Time Frame: Baseline and the efficacy assessment phase (Week 20 to Week 27)
Population: Full analysis set participants with observed data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 237 | 227
percent change | 0.58 (0.29) | -6.69 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p < 0.001, Repeated Measures Mixed Effects Model; [statistical method as in outcome 3, analysis 1]; Mean Difference = -7.20, 95% CI 2-sided [-8.38 to -6.03], Standard Error of Mean 0.60 — Etelcalcetide - Placebo

5. Secondary Outcome: Percent Change From Baseline in Predialysis Corrected Calcium Phosphorus Product (cCa x P) During the Efficacy Assessment Phase
Time Frame: Baseline and the efficacy assessment phase (Week 20 to Week 27)
Population: Full analysis set participants with observed data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 234 | 223
percent change | -1.06 (1.42) | -15.84 (1.57)
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p < 0.001, Repeated Measures Mixed Effects Model; [statistical method as in outcome 3, analysis 1]; Mean Difference = -14.58, 95% CI 2-sided [-18.65 to -10.51], Standard Error of Mean 2.07 — Etelcalcetide - Placebo

6. Secondary Outcome: Percent Change From Baseline in Predialysis Phosphorus During the Efficacy Assessment Phase
Time Frame: Baseline and the efficacy assessment phase (Week 20 to Week 27)
Population: Full analysis set participants with observed data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 234 | 223
percent change | -1.60 (1.42) | -9.63 (1.61)
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p < 0.001, Repeated Measures Mixed Effects Model; [statistical method as in outcome 3, analysis 1]; Mean Difference = -8.04, 95% CI 2-sided [-12.15 to -3.92], Standard Error of Mean 2.09 — Etelcalcetide - Placebo

ADVERSE EVENTS:
Time Frame: From Day 1 until 30 days after the last dose; the treatment period was 26 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Etelcalcetide
Serious Adverse Events (participants affected / at risk) | 71/259 | 62/252
Other Adverse Events (participants affected / at risk) | 132/259 | 199/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | Etelcalcetide (N=252)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 3
Angina pectoris (Cardiac disorders) | 2 | 1
Angina unstable (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 4 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Primary hyperaldosteronism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Catheter site haematoma (General disorders) | 0 | 1
Hernia obstructive (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 0 | 3
Sudden death (General disorders) | 1 | 1
Surgical failure (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arteriovenous fistula site infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Burn infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile sepsis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Herpes zoster meningoencephalitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 3 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 4
Postoperative abscess (Infections and infestations) | 1 | 0
Prostatic abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Sepsis syndrome (Infections and infestations) | 1 | 0
Skin graft infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral myocarditis (Infections and infestations) | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 2
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Graft complication (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1
Skin graft failure (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 4 | 2
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 6
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2
Obesity (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 2 | 1
Dementia (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hyperglycaemic seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 2 | 0
Uraemic encephalopathy (Nervous system disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Palpable purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Finger amputation (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Poor peripheral circulation (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Venous stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | Etelcalcetide (N=252)
Anaemia (Blood and lymphatic system disorders) | 13 | 8
Diarrhoea (Gastrointestinal disorders) | 25 | 35
Nausea (Gastrointestinal disorders) | 18 | 23
Vomiting (Gastrointestinal disorders) | 8 | 19
Upper respiratory tract infection (Infections and infestations) | 15 | 13
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 12 | 16
Blood calcium decreased (Investigations) | 31 | 168
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 28
Headache (Nervous system disorders) | 11 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 10
Hypertension (Vascular disorders) | 12 | 18
Hypotension (Vascular disorders) | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.